CLINICAL TRIAL: NCT04023773
Title: Assess Safety and Feasibility of Sequential Hypothermic Oxygenated Machine Perfusion and Normothermic Machine Perfusion to Preserve Extended Criteria Donor Livers for Transplantation
Brief Title: Sequential Hypo- and Normo-thermic Perfusion to Preserve Extended Criteria Donor Livers for Transplantation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koji Hashimoto (Other)
Responsible Party: Sponsor-Investigator, Koji Hashimoto, Staff Physician, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sequential perfusion
Record Dates: First submitted 2019-07-10; First posted 2019-07-18 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Intervention Model Description: Eighteen extended criteria donor livers will be transplanted after receiving sequential hypothermic and normothermic machine perfusion preservation prior to transplantation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Liver perfusion (Experimental): Device: Liver Machine Perfusion (MP) Device
  The liver grafts will be preserved at hypothermic and normothermic temperature on the institutional-developed Liver MP Device, and have continuous perfusion with oxygen supply in the ex vivo organ preservation phase.
  Interventions: Device: Liver Machine Perfusion (MP) device

INTERVENTIONS:
Device: Liver Machine Perfusion (MP) device — Donor livers will have ex vivo continuous perfusion on the institutional-developed Liver MP device. The temperature of liver grafts will be controlled during perfusion.

SUMMARY:
Hypothermic machine perfusion (HMP) has been shown to be beneficial to preserve extended criteria donor (ECD) livers for transplantation. Normothermic machine perfusion (NMP) had the same benefits and also the convenience on liver quality assessment. The investigators proposed to do sequential HMP (1-4 hours) and NMP (1-14 hours) on 18 ECD transplanted human livers by using an institutional-developed perfusion device for liver transplantation.

DETAILED DESCRIPTION:
Liver transplantation is a successful therapy on the patients with end-stage liver disease, however is limited by the shortage of donor organs. Donor criteria were expanded in the past decades, however the extended criteria donor (ECD) livers may induce a higher risk of complications. Static cold storage (SCS) is the standard procedure for ex vivo liver preservation for about 4 decades, but has the limitation on preserving ECD livers and especially the inconvenience to evaluate liver quality prior to transplantation. Hypothermic (4-8 Celsius degree) machine perfusion (HMP) and Normothermic (35-37 Celsius degree) machine perfusion (NMP) have been shown to be beneficial to preserve extended criteria donor (ECD) livers respectively. NMP also had the convenience on liver quality assessment. The investigators had an institutional-developed device for liver NMP used on 25 patients with the FDA's IDE approval. In the present study the investigators are proposing to expand the use of the device on sequential HMP (1-4 hours) and NMP (1-14 hours) on 18 ECD transplanted human livers. This will be a single center prospective pilot study. The liver metabolism and hydrodynamics during perfusion will be recorded. The transplant procedure and post-transplant care will follow the clinical standard of care. The follow-up period is 12 months after transplantation. The primary end point will be the rate of patient survival and primary non function (PNF) within 30 days after transplantation, while the secondary end points will be: Early Allograft Dysfunction (EAD), 6 months patient and graft survival, peak liver function tests in the first 7 days after transplantation, surgical outcomes (operative time, transfusion requirement etc.), rate of post-transplant kidney failure, assessment of histological ischemia reperfusion (liver and bile duct), rate of vascular complications, rate of biliary complications, hospital and ICU length of stay, rejection rate, infection rate, the ability to predict function based on "on-pump" viability markers, and the incidence of adverse effect (AE).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing liver transplantation
* Age 18 or older at the time of transplantation
* Willingness and ability to comply with the study procedures
* Signed Informed Consent Form

Exclusion Criteria:

* Recipient of partial grafts (split and living donors)
* Mentally or legally incapacitated subjects
* Inability to understand the procedures due to language barriers
* Multiorgan transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
patient survival at 1 month post-transplant | 1 month post-transplant
  Patient survival will be recorded at 1 month post transplantation.
graft survival at 1 month post-transplant | 1 month post-transplant
  graft survival will be recorded at 1 month post transplantation. The allograft will be considered lost if a patient has a primary non function (PNF), liver re-transplant or in the event of patient death.

SECONDARY OUTCOMES:
rate of post-transplant early allograft dysfunction (EAD) | in the first 7 days after transplantation
  EAD is defined as the presence of one or more of the following previously defined postoperative laboratory analyses reflective of liver injury and function: bilirubin ≥10mg/dL on post-operative day (POD) 7, international normalized ratio (INR) ≥1.6 on POD 7, and alanine or aspartate aminotransferases (ALT or AST) >2000 IU/L within the first 7 days.
patient survival at 6 month post-transplant | 6 month post-transplant
  patient survival will be recorded at 6 months post transplantation.
graft survival at 6 month post-transplant | 6 month post-transplant
  graft survival will be recorded at 6 month post transplantation. The allograft will be considered lost if a patient has a primary non function (PNF), liver re-transplant or in the event of patient death.
Estimated blood loss at transplant surgery | during surgery
  Estimated blood loss (ml) during transplant surgery
peak alanine aminotransferases in the first 7 days after transplantation | in the first 7 days after transplantation
  peak level (U/L) of alanine aminotransferases in the first 7 days after transplantation
peak aspartate aminotransferases in the first 7 days after transplantation | in the first 7 days after transplantation
  peak level (U/L) of aspartate aminotransferases in the first 7 days after transplantation
total bilirubin on post-operative day 7 | on post-operative day 7
  total bilirubin (mg/dL) on post-operative day 7
international normalized ratio on post-operative day 7 | on post-operative day 7
  international normalized ratio on post-operative day 7
Hospital length of stay | up to 36 weeks
  Length of stay (days) in the hospital at the time for transplantation
ICU length of stay | up to 36weeks
  Length of stay (days) in ICU at the time after liver transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Koji Hashimoto, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No